CLINICAL TRIAL: NCT05683886
Title: A Single-arm, Open, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of KC1036 in the Patients with Advanced Recurrent or Metastatic Thymic Tumors
Brief Title: A Study of KC1036 in Patients with Advanced Thymic Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC1036-II-02
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Thymic Tumors
MeSH Terms: conditions — Thymus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KC1036 (Experimental): 60mg QD
  Interventions: Drug: KC1036

INTERVENTIONS:
Drug: KC1036 — Patients take 60mg QD of KC1036 for the efficacy and safety study. KC1036 are given orally once daily, 21 days as a cycle.

SUMMARY:
This is a single arm，open-label, multicentric, phase II study to evaluate the efficacy and safety of KC1036 in patients with advanced recurrent or metastatic thymoma or thymic carcinoma.

DETAILED DESCRIPTION:
Thymus tumor is a relatively rare type of thoracic tumor. Patients with thymus tumor who have failed to receive first-line chemotherapy lack of effective therapeutic drugs and clinical need is urgent. Previous phase I study showed that KC1036 has a good therapeutic effect in patients with advanced thymic tumors, and KC1036 is safe and well tolerated in patients with advanced tumors. This study further explored the efficacy and safety of KC1036 in patients with advanced thymic tumors.

Patients will receive continuous treatment with oral KC1036 60 mg once daily. Each cycle will be considered as 21 days of treatment; safety was assessed every 21 days. Tumor assessement will be done every two cycles. Treatment should be administered until documented disease progression, unacceptable toxicity, or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thymoma or thymic carcinoma confirmed by cytologically or histologically (WHO Classification of Thoracic Tumors 5th ed), including all pathological subtypes;
* Patients with advanced recurrent, unresectable and/or metastatic thymic tumor as defined by the Masaoka-Koga stage;
* Subsequent relapse of disease following first-line systemic chemotherapy;
* Patients with at least one measurable lesion as defined by RECIST V1.1; Measurable lesions located within the radiation field of previous radiotherapy or after local treatment can also be selected as target lesions if progression is confirmed.
* Eastern Cooperative Oncology Group performance status score of 0 or 1;
* Life expectancy > 12 weeks;
* Adequate organ and marrow function;
* Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* Patients with thymus neuroendocrine tumors;
* Any patient who is known to have central nervous system (CNS) metastasis or imaging shows a risk of CNS metastasis;
* Previous (within the last 5 years) or current malignancies at other sites;
* Gastrointestinal abnormalities;
* Cardiovascular and cerebrovascular diseases;
* Patients who have previous treatment with small molecule VEGFR-TKI (except patients whose treatment cycle is less than 2 weeks due to intolerance or other reasons); Patients who have previous treatment with PD-1 / PD-L1 antibody combined with small molecule VEGFR-TKI;
* Involved in other clinical trials within 4 weeks before enrollment; Prior anti-tumor therapies with chemotherapy, cytotherapy, immunotherapy, operation (Interventional therapy excepted) within 4 weeks 4 weeks before enrollment; Prior radiotherapy (palliative radiotherapy excepted) within 2 weeks; Prior small-molecule targeted therapy within 2 weeks or 5 half-lives.
* Presence of unresolved toxicities from prior anti-tumor therapy, defined as having not resolved to NCI CTCAE V5.0 grade 0 or 1 with the exception of alopecia;
* Skin wound, surgical site, wound site, mucous membrane severe ulcer or fracture comfirmed as having not recovered;
* Uncontrolled mass pleural effusion, ascites, and pericardial effusion;
* Active autoimmune diseases: Myasthenia gravis, pure red cell aplastic anemia, systemic lupus erythematosus, inflammatory bowel disease, etc;
* Need immunosuppressive agents or hormone therapy for immunosuppression, , and still need immunosuppressive therapy within 2 weeks before enrollment;
* Active bacterial, viral or fungal infection; Fever of unknown cause (> 38.5℃) occurred within 2 weeks before enrollment;
* Patients who are positive for both Hepatitis B surface antigen (HBsAg) and hepatitis B virus deoxyribonucleic acid (HBV-DNA) quantification results; Patients who are positive for both hepatitis C virus antibody (HCAB) and hepatitis C virusribonucleic acid (HCV-RNA) quantification results; Patients who are positive for human immunodeficiency virus (HIV);
* Pregnant or lactating women;
* Patients who do not take contraception during the study period and within 6 months after the study;
* Patients with insufficient compliance as evaluated by investigator;
* The investigator believes that it is not suitable to patient in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | approximately 2 year
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | approximately 2 year
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | approximately 2 year
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | approximately 2 year.
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.
Adverse events (AEs) | approximately of 2 year
  Incidence of treatment-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Ph.D, Principal Investigator — West China Hospital; Wentao Fang, Ph.D, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No